CLINICAL TRIAL: NCT00714896
Title: A Stepped-Care Intervention for Current and Former Smokers in Outpatient Chemical Dependency Treatment
Brief Title: Interventions for Smoking Among Persons in Recovery
Acronym: INSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kaiser Permanente (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Janice Tsoh, Ph.D., Associate Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P50DA009253-14-DevStudy2; H10315-28247-03; P50DA009253-14 (NIH)
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; nicotine dependence; stage-based intervention; nicotine replacement medications; counseling; substance abuse treatment
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Assessment only + referral list to State quitline and smoking cessation education classes at Kaiser
  Interventions: Behavioral: Control
- 2 (Experimental): Participants will receive self-help information handouts, expert system intervention that includes a stage-based manual and individualized written feedback reports plus in-person brief stage-appropriate counseling at baseline and 3-month assessment. Current smokers who indicate desire to quit smoking or former smokers who indicate high cravings for cigarettes will be offered nicotine replacement medications. Participants will receive three telephone counseling sessions delivered between baseline and 3 month at weeks 2, 4 and 8. As-needed telephone check-calls will be provided to participants on and 2 days after quit date, or to participants who have quit smoking and anticipate high risk situations.
  Interventions: Behavioral: Stepped-Care

INTERVENTIONS:
Behavioral: Stepped-Care — * stage-based expert system written intervention at baseline and 3 months
  * in-person stage appropriate counseling at baseline and 3 months
  * telephone counseling sessions at weeks 2,4 and 8,
  * as-needed brief check-in calls on or 2 days after quit date for those who have set a quit date; and/or check-in calls on days with anticipated high risk situations for former smokers or those who have quit smoking during the study
  * optional NRT nicotine replacement therapy in the forms of patch, gum or lozenge for current smokers who are ready to quit smoking and/or for former smokers who report significantly strong smoking urges
  Arms: 2
Behavioral: Control — Referral list to smoking cessation classes at Kaiser and the California Smokers Helpline
  Arms: 1

SUMMARY:
Examine the efficacy of a stepped-care smoking cessation intervention for current and former smokers in chemical dependency treatment programs. We hypothesize that those who received the stepped-care intervention will be more likely to report smoking abstinence and drug or alcohol abstinence at 6 months.

DETAILED DESCRIPTION:
The objective of the study is to document and systematically investigate the use of smoking cessation strategies targeting substance abuse outpatient smokers at various level of readiness to quit smoking. Little is known regarding the best practices in treating tobacco use among clients in drug abuse treatment and very few drug abuse treatment programs currently offer smoking cessation services. The purpose of this developmental study is to develop and pre-test a stepped-care smoking cessation intervention in an outpatient drug abuse treatment program at a managed care setting that targets both current and former smokers. The stepped-care intervention consists of various components that aim at matching the treatment needs of smokers across the whole spectrum of smoking status and readiness to quit smoking. The following specific aims will be pursued:

1. Develop a stepped-care smoking cessation intervention targeting both current and former smokers who are admitted to an outpatient drug abuse treatment program. Special attention will be paid to former smokers, as intervention techniques for them are not well developed. Also, intervention content will be modified from that used in smoking interventions with the general population to content that is targeted at smokers who are in drug abuse treatment
2. Pre-test the efficacy of the stepped-care smoking cessation intervention.
3. Examine the feasibility of implementing the stepped-care smoking cessation intervention.
4. Examine the impact of the smoking intervention on drug and alcohol use outcomes at 6-month post initiation of smoking cessation treatment.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* over the age of 18
* currently enrolled in outpatient treatment program for drug and/or alcohol use and have received minimally 30 days of continuous treatment for drug and/alcohol in any outpatient treatment program(s) for drug and/or alcohol use for at least one month
* have regularly smoked cigarettes for at least one year in their lifetime
* have smoked within the past 5 years

Exclusion Criteria:

* clients with a life-threatening disease
* currently at imminent risk of committing suicide, or currently pregnant
* currently in treatment for nicotine dependence elsewhere
* cannot be reached by telephone (unable to provide a phone number where the participant can be reached directly
* non-English speakers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
CO verified self-report 7-day smoking abstinence prior to assessment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Janice Tsoh, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Kaiser Permanente Central Diablo (Wlanut Creek/ Martinez), Walnut Creek, California, United States